CLINICAL TRIAL: NCT05488821
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of the Oral Pan-RAF Inhibitor QLH11906 in Subjects With Advanced Solid Tumors Harboring MAPK Pathway Alterations.
Brief Title: Safety, Tolerability and Pharmacokinetics Study of QLH11906 in Patients With Advanced Solid Tumors Harboring MAPK Pathway Alterations.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLH11906-101
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumors Harboring MAPK Pathway Alterations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLH11906 (Experimental): QLH11906 Tablets
  Interventions: Drug: QLH11906

INTERVENTIONS:
Drug: QLH11906 — QLH11906 only

SUMMARY:
This is an open label, phase 1 clinical study to evaluate the safety and tolerability of different doses of QLH11906 monotherapy in patients with relapsed/refractory, unresectable locally advanced or metastatic advanced solid tumors with abnormal MAPK pathway, and determine the Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD, if MTD cannot be determined) and Recommended Dose in Phase II Clinical Studies (Recommended Phase II Dose, RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. The subjects participated voluntarily, signed the informed consent, and were able to abide by the research procedures.
2. Subjects with advanced (metastatic or unresectable) solid tumors with histologically confirmed MAPK signaling pathway alteration.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
4. Subjects are able to swallow and retain oral medication without any clinically significant gastrointestinal abnormalities that alter absorption.
5. Subjects (including women and men) agree to use effective contraception for contraception from the time of signing the informed consent form to 180 days after the last use of the study drug. Female subjects of childbearing age cannot be pregnant or breastfeeding.

Exclusion Criteria:

1. Subjects received systemic anticancer therapy within 2 weeks prior to the first dose.
2. Subjects received radical radiotherapy within 4 weeks before the first administration, or received local palliative radiotherapy for bone metastases within 1 week.
3. Subjects who have received inhibitors or inducers of CYP3A4 within 1 week before the first dose; or within 5 half-lives of the drug; or subjects who need to continue to receive these drugs during the study period.
4. Active bacterial, fungal, or viral infection requiring systemic therapy within 1 week prior to the first dose.
5. Subjects with symptomatic central nervous system (CNS) metastases and/or cancerous meningitis.
6. Cardiovascular and cerebrovascular diseases with clinical significance.
7. Clinically uncontrollable serous effusion (eg, pleural effusion that cannot be controlled by drainage or other methods).
8. Active gastrointestinal disease or other conditions that significantly interfere with drug absorption.
9. Known immediate or delayed hypersensitivity reactions or idiosyncratic reactions to the investigational treatment-related chemotherapeutic drugs and their excipients.
10. Human immunodeficiency virus (HIV) positive test result and Treponema pallidum antibody positive.
11. Hepatitis B virus surface antigen (HBsAg) positive and viral deoxyribonucleic acid (HBV DNA) > 2000 IU/ml or 104 copies/ml (only the centers that can perform qualitative examination, the HBV DNA test result is positive or high detection limit); hepatitis C virus antibody positive and viral ribonucleic acid (HCV RNA) positive.
12. Other malignant tumors occurred within 2 years before study enrollment. (Except: Bowen's disease; cured basal cell or squamous cell skin cancer; prostate cancer with a Gleason score of 6; treated cervical carcinoma in situ.)
13. Pregnant or lactating women.
14. Any pre-existing serious or unstable disease (except for the above-mentioned malignant tumors), mental disease or any disease or medical condition that the investigator considers may interfere with the subject's safety, obtaining informed consent, or complying with research procedures.
15. Concurrent participation in other clinical trials using experimental therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
MTD/MAD | Up to 24 approximately months
  The Maximum Tolerated Dose (MTD) will be determined during dose escalation using a Bayesian Optimal Interval (BOIN) design.The maximum administrated dose (MAD) is defined as the highest dose of all groups if MTD can not be determined.
RP2D | Up to 24 approximately months
  Recommended dose for phase II trials

SECONDARY OUTCOMES:
Adverse Events (AEs) /Serious Adverse Events (SAEs) | Up to 24 approximately months
Area under the concentration-time curve（AUC） | Up to 24 approximately months
  Pharmacokinetic (PK) parameters of QLH11906 monotherapy, including Area under the concentration-time curve（AUC）
Overall response rate (ORR) | Up to 24 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria, including objective response rate(ORR).
Duration of response (DoR) | Up to 24 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria, including duration of response(DOR).
Disease control rate (DCR) | Up to 24 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria, including disease control rate(DCR).
Maximum concentration (Cmax) | Up to 24 approximately months
  Pharmacokinetic (PK) of QLH11906 monotherapy, including Maximum concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital, Shandong, China